CLINICAL TRIAL: NCT00233558
Title: Multicentre, Randomised, Open Label Study Comparing a "Scheduled Steroid Reduction Strategy" Versus a Free Steroid Reduction Strategy (Physician's Usual Practice for Reducing Steroids) in Patients With Active RA Treated With Humira 40 mg Eow + MTX During 9 Months
Brief Title: Open-Label Steroid Reduction Study of Adalimumab With Methotrexate in Patients With Active Rheumatoid Arthritis
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Study terminated due to low subject enrollment. Safety results consistent with product label.
Sponsor: Abbott (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FRAN-04-002
Record Dates: First submitted 2005-09-13; First posted 2005-10-06 (Estimated); Last update posted 2007-04-24 (Estimated); Status verified 2007-04

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Adalimumab; Methotrexate

INTERVENTIONS:
Drug: adalimumab (up to 9 months exposure)
Drug: methotrexate

SUMMARY:
The purpose of the study is to evaluate the clinical efficacy of scheduled versus free reduction of steroid treatment in patients with active RA treated with adalimumab + MTX

ELIGIBILITY:
Inclusion Criteria:

* Subject is age 18 or older and in good health (Investigator discretion) with a recent stable medical history
* Subject has a diagnosis of rheumatoid arthritis as defined by the 1987-revised ACR criteria

Exclusion Criteria:

* Subject considered by the investigator, for any reason, to be an unsuitable candidate for the study
* Female subject who is pregnant or breast-feeding or considering becoming pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160
Dates: Start 2005-06

PRIMARY OUTCOMES:
Corticoid reduction and DAS 28

SECONDARY OUTCOMES:
Patient reported outcomes
Clinical response indicators
Safety parameters

CONTACTS AND LOCATIONS:
Overall Officials: Global Medical Information, Study Director — Abbott
Locations (1):
- Global Medical Information - Abbott, North Chicago, Illinois, United States